CLINICAL TRIAL: NCT05403853
Title: A Performance Evaluation of the LumiraDx Point of Care HbA1c Device
Acronym: PHADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LumiraDx UK Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S-CLIN-PROT-00009
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: IVD Performance Evaluation Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monitoring of Diabetes Mellitus (Experimental): Venous blood draw of up to 24ml and up to 4 fingersticks
  Interventions: Diagnostic Test: Venepuncture; Diagnostic Test: Fingerstick

INTERVENTIONS:
Diagnostic Test: Venepuncture — Venous blood draw
Diagnostic Test: Fingerstick — Capillary Blood Draw

SUMMARY:
In patients who have diabetes, symptoms of diabetes or attending a diabetic clinic the study will evaluate agreement between the HbA1c measurements from the LumiraDx POC HbA1c assay and the Tosoh G8, as an aid in the monitoring of diabetes Mellitus

DETAILED DESCRIPTION:
This is a performance evaluation study designed to assess the precision and accuracy of the LumiraDx Point of Care (POC) HbA1c test when used in patients presenting for assessment or monitoring of diabetes.

The LumiraDx POC HbA1c test is a quantitative immunoassay providing results near to the patient in under 10 minutes. The accuracy of the LumiraDx POC HbA1c test will be assessed using capillary whole blood, and venous blood, by comparison to the HbA1c results obtained from the same individuals as analysed by trained laboratory professionals using a CE marked laboratory reference device.

The results of this study are intended to be used for regulatory filings for use as an in vitro diagnostic test in the UK, European Union (EU) and other relevant geographies.

Adult males and females attending out-patient, community diabetes and research clinics for HbA1c measurements will be included in the study. Subjects may also be invited to take part via the diabetes research register or by invitation from independent clinical research sites. All subjects recruited will be willing and able to give written informed consent. Approximately 400 subjects will be recruited to ensure that sufficient suitable subjects are enrolled and to allow for a small level of exclusions. The power calculation requires a minimum of 360 valid subjects in total.

After obtaining written informed consent, up to 24mL of venous blood will be obtained from venepuncture into anticoagulated blood tubes. Capillary blood samples should be collected via fingerstick. Finger stick blood should be collected using the transfer loop and placed in the sample tube before addition to the strip for immediate measurement of HbA1c on the LumiraDx POC instrument (one after the other).

Of the drawn blood tubes, one tube is used immediately with the LumiraDx POC HbA1c test. To do this, the clinical staff member lyses a small sample using the lysis kit and then places the sample on the Test Strip which has already been inserted into the LumiraDx POC Instrument. After approx. 8 minutes, the result is displayed on the screen.

The HbA1c results obtained will be used in a set of comparative analyses designed to determine the performance characteristics of the LumiraDx HbA1c test. This study is an observational, cross-sectional design. As an observational study of an investigative device, results obtained during the course of the study will not inform or alter patient management or treatment decisions in any way.

ELIGIBILITY:
Inclusion Criteria:

* Subject greater that 18 years of age
* Willing and able to provide written informed consent and comply with study procedures
* Presenting at clinic for assessment of diabetes, diagnosis of diabetes or HbA1c monitoring of diabetes therapy, or attending an independent research clinic or present on a diabetes research database.

Exclusion Criteria:

* Patient has previously participated in this study
* Investigator opinion of short life expectancy of < 1 month
* Patients who have received an Investigational Medicinal Product within the last 30 days
* Haemodynamically unstable (e.g. cardiogenic shock)
* Conditions where HbA1c cannot be used for diagnosis (see John et al., 2011 (4). Pregnancy or two months postpartum, patients with symptoms of diabetes for less than two months, patients at high diabetes risk who are acutely ill, patients taking medication that can cause a rapid glucose rise such as corticosteroids, antipsychotic drugs (2 months or less); acute pancreatic damage including pancreatic surgery, renal failure, HIV infection or patients who have received a blood transfusion or cancer chemotherapy within 3 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
Performance of the LumiraDx POC HbA1c assay when compared to a current CE marked reference method in patients being assessed for diagnosis or monitored for diabetes. | 2 months
  Measurement of blood samples from participants who have been diagnosed with diabetes mellitus or who are being monitored for symptoms of diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Rory McCrimmon, Principal Investigator — NHS Tayside; Isabel Howat, Principal Investigator — NHS Lanarkshire; Catherine Patterson, Principal Investigator — NHS Fife; Louise Brown, Principal Investigator — Intelligent Clinical
Locations (4):
- United Kingdom (4):
  - Ninewells Hospital, Dundee, Dundee
  - Intelligent Clinical, Glasgow
  - NHS Lanarkshire, Glasgow
  - Victoria Hospital, Kirkcaldy

IPD SHARING:
Plan to Share IPD: No